CLINICAL TRIAL: NCT05835999
Title: Clinical Evaluation of mTORC1 Inhibition for Geroprotection
Brief Title: Everolimus Aging Study
Acronym: EVERLAST
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-1519; 1U01AG076941-01 (NIH); A534255 (Other: UW Madison); Protocol Version 4/30/2025 (Other: UW Madison)
Record Dates: First submitted 2023-04-03; First posted 2023-05-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Aging; Insulin Resistance
Keywords: rapamycin; rapamycin analog; mTOR; everolimus
MeSH Terms: conditions — Insulin Resistance | interventions — Everolimus

STUDY DESIGN:
Intervention Model Description: This is a randomized, placebo-controlled, double-blind, 24-week clinical trial using everolimus in middle-aged to older adults. This study will follow a "double-dummy" design where participants will be randomized 1:1:1 in a double-blinded fashion to one of three groups: 1) everolimus once daily (0.5 mg/day) plus placebo once weekly, 2) placebo once daily plus everolimus once weekly (5mg/week) or 3) placebo once daily and placebo once weekly. The double dummy design preserves the double-blind for both placebo versus everolimus and for daily versus weekly dosing schedules. Everolimus and placebo will be over encapsulated to be indistinguishable from one another.
  There will also be a group of young, healthy individuals who will complete baseline testing only and not the intervention. This group allows the determination if everolimus changes any molecular and physiological outcomes in older adults toward that of a young, healthy reference group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Daily Everolimus (0.5 mg/day) and Weekly Placebo (Experimental): Once daily (0.5 mg) everolimus and once weekly placebo taken orally for 24 weeks
  Interventions: Drug: Everolimus 0.5 MG once per day; Drug: Placebo once per week
- Daily Placebo and Weekly Everolimus (5mg/week) (Experimental): Once daily placebo and once weekly (5 mg) everolimus taken orally for 24 weeks
  Interventions: Drug: Everolimus 5 MG once per week; Drug: Placebo once per day
- Daily Placebo and Weekly Placebo (Placebo Comparator): Once daily placebo and once weekly placebo taken orally for 24 weeks
  Interventions: Drug: Placebo once per day; Drug: Placebo once per week
- Young Adult Reference Group (No Intervention): Baseline testing only

INTERVENTIONS:
Drug: Everolimus 0.5 MG once per day — Everolimus is considered an mTOR kinase inhibitor
  Arms: Daily Everolimus (0.5 mg/day) and Weekly Placebo
Drug: Everolimus 5 MG once per week — Everolimus is considered an mTOR kinase inhibitor
  Arms: Daily Placebo and Weekly Everolimus (5mg/week)
Drug: Placebo once per day — No therapeutic effect
  Arms: Daily Placebo and Weekly Everolimus (5mg/week); Daily Placebo and Weekly Placebo
Drug: Placebo once per week — No therapeutic effect
  Arms: Daily Everolimus (0.5 mg/day) and Weekly Placebo; Daily Placebo and Weekly Placebo

SUMMARY:
The objective of this project is to determine if mTORC1 inhibition by 24 weeks of daily (0.5 mg/day) or weekly (5 mg/week) everolimus can safely improve physiological and molecular hallmarks of aging in humans. Participants who are 55-80 years old and insulin resistant or prediabetic will be randomized to treatment and can expect to be on study for up to approximately 38 weeks. Participants aged 18-35 will not receive the intervention and can expect to be on study for up to approximately 8 weeks.

DETAILED DESCRIPTION:
Pharmacological inhibition of mechanistic target of rapamycin (mTOR) has been repeatedly demonstrated to extend lifespan and prevent or delay several age-related diseases in diverse model systems. However, the risk of potentially serious side effects in humans have thus far prevented the long-term use of the mTOR inhibitor rapamycin as a therapy for aging and age-related diseases. Therefore, it remains unknown whether rapamycin or rapamycin analogs (rapalogs) can safely improve healthy aging in humans.

The objective of this project is to determine if 24 weeks of daily low dose (0.5 mg/day) or weekly intermittent (5 mg/week) treatment with the rapalog everolimus can safely improve physiological and molecular hallmarks of aging in middle-aged to older insulin resistant adults who are at high risk for nearly every age-related condition.

Using a double-blinded, randomized, placebo-controlled clinical trial, the investigators will perform a battery of gold-standard and innovative techniques to test the hypothesis that daily low dose or weekly everolimus treatment will improve 4 inter-related domains of physiological aging: metabolic, cardiac, cognitive, and physical function. The investigators will also assess the incidence of adverse events and changes from baseline blood chemistry, blood cell counts, lipids, glucose, and insulin.

To comprehensively examine the molecular target specificity and the impact on mechanisms of aging by everolimus, the team will evaluate mTORC1 and mTORC2 signaling, assess mitochondrial bioenergetics, and perform a multi-omics approach (epigenomics, transcriptomics, proteomics, lipidomics, and metabolomics) in blood and/or muscle biopsy samples.

ELIGIBILITY:
Inclusion Criteria: Adults aged 55-80 years old

* Free of overt chronic disease
* Willing to provide informed consent
* Willing to comply with all study procedures and be available for the duration of the study
* Able to use and be contacted by the telephone
* Ability to take oral medication
* Insulin Resistant defined by HOMA-IR greater than or equal to 1.5 or prediabetic defined as:

  * impaired fasting glucose (100-125 mg/dL)
  * HbA1c (5.7-6.4 percent)
  * glucose 2 hours after a 75 gram oral glucose tolerance test (140-199 mg/dL)
  * previous diagnosis of prediabetes in the past year
* Not planning to change diet or physical activity status
* Adequate organ function as indicated by standard laboratory tests: hematology (complete blood count), clinical chemistry and urinalysis
* Females of childbearing potential must have a negative urine pregnancy test before DEXA and before the oral glucose tolerance test (OGTT). A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Women of childbearing potential in sexual relationships with men must use an acceptable method of contraception from 30 days prior to enrollment until 4 weeks after completing study visits. Males must agree to avoid impregnation of women during and for four weeks after completing study visits through use of an acceptable method of contraception.

  * Note: Includes, but is not limited to, barrier with additional spermicidal foam or jelly, intrauterine device, hormonal contraception (started at least 30 days prior to study enrollment), intercourse with men who underwent vasectomy.

Inclusion Criteria: Younger Adults aged 18-35 (No intervention)

* Free overt chronic disease

Exclusion Criteria:

* Pregnancy or breastfeeding
* Heart disease
* Cerebrovascular disease
* Cancer or less than 5 years in remission
* Chronic respiratory disease
* Chronic liver disease
* Diabetes
* Alzheimer's
* Chronic kidney disease
* For those undergoing muscle biopsy: problems with bleeding, on medication that prolongs bleeding time
* Taking azathioprine (Imuran), cyclosporine (Gengraf, Neoral, Sandimmune), dexamethasone (Decadron, Dexpak), methotrexate (Rheumatrex, Trexall), prednisolone (Orapred, Pediapred, Prelone), prednisone (Sterapred), sirolimus (Rapamune), and tacrolimus (Prograf) or other medications proposed to lower the immune system. Daily use of high potency topical corticosteroids used on greater than or equal to 10% of body surface area will not be eligible. Nasal sprays or inhaled corticosteroids will be reviewed on a case-by-case basis.
* Taking strong or moderate CYP3A4 and/or P-glycoprotein (PgP) inhibitors
* Taking strong CYP3A4 activators
* Taking daily NSAIDs with the exception of baby asprin (81 mg)
* Subjects who are not willing to restrict the use of grapefruit, grapefruit juice, and other foods that are known to inhibit cytochrome P450 and PgP activity and may increase everolimus exposures and should be avoided during treatment
* Subjects who are not willing to restrict the use of St. John's Wort (Hypericum perforatum) because it may decrease everolimus exposure unpredictably
* Subjects who are not willing to avoid blood donations 8 weeks prior to the first visit and 8 weeks after the last visit
* For those undergoing MRI, contraindications with MRI which could include metal on your body
* Low white-blood cell count (<4,000 cell/µL)
* History of stomatitis or ulcers in the mouth
* Those on glucose lowering drugs
* Participating in intensive exercise training program (high to moderate intensity exercise greater than 150 minutes per week) or planning to start new exercise program during study period
* Tobacco use
* Allergies to lidocaine or everolimus
* Subjects currently enrolled in other clinical trials. Subjects may be eligible after a washout period that will be reviewed on a case by case basis.
* Individuals with limited English proficiency
* Subjects who are planning to have elective surgery 12 weeks prior to or during the intervention

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Metabolic Function: Change in peripheral insulin sensitivity | 0 (pre-intervention) and 24 weeks (post-intervention)
  Change (pre to post) in peripheral insulin sensitivity measured by glucose disposal rate relative to circulating insulin during a dual tracer 75g oral glucose tolerance test (OGTT).

SECONDARY OUTCOMES:
Cardiac Function: Change in fractional shortening velocity | 0 (pre-intervention) and 24 weeks (post-intervention)
  Cardiac Function will be assessed by measuring the change in fractional shortening velocity determined during the echocardiogram.
Cognitive Function: Change in cerebral blood flow | 0 (pre-intervention) and 24 weeks (post-intervention)
  Change in blood flow in posterior cingulate, medial temporal lobe (hippocampus and parahippocampus) and inferior frontal cortex assessed by brain MRI (4D Flow, Arterial Spin Labeling).
Safety: Number of Participants with Adverse Events | up to 36 weeks
  Safety will be measured in part by reporting the number of participants with adverse events.
Safety: Change in concentration of blood metabolites/enzymes | 0 (pre-intervention), 4, 8, 12, 16, 20, and 24 weeks (post-intervention)
  Safety will be measured in part by reporting the change in the blood concentration of metabolites and enzymes as assessed by a complete metabolic panel
Safety: Changes in concentration of blood lipids | 0 (pre-intervention), 4, 8, 12, 16, 20, and 24 weeks (post-intervention)
  Safety will be measured in part by reporting the changes in the concentration of blood lipids.
Safety: Changes in number of blood cells | 0 (pre-intervention), 4, 8, 12, 16, 20, and 24 weeks (post-intervention)
  Safety will be measured in part by reporting the changes in the number of blood cells as determined by blood cell count with differential
Safety: Changes in HbA1c (%) | pre-intervention baseline, post-intervention up to 24 weeks
  Safety will be measured in part by reporting the changes in the percentage of glycosylated hemoglobin (Hba1c (%))
Safety: Changes in concentration of insulin | 0 (pre-intervention), 4, 8, 12, 16, 20, and 24 weeks (post-intervention)
  Safety will be measured in part by reporting the changes in fasting blood insulin concentration
mTOR signaling: Change in phosphorylation of downstream targets of mTOR complex 1 and complex 2 as assessed by immunoblotting and immunoprecipitation. | pre-intervention baseline, post-intervention up to 24 weeks
  mTOR signaling will be assessed by measuring the change in phosphorylation of downstream targets of mTOR complex 1 and complex 2 via immunoblotting in muscle and/or peripheral mononuclear blood cells (PMBCs).

OTHER OUTCOMES:
Physical Function: Change in cardiorespiratory fitness | 0 (pre-intervention) and 24 weeks (post-intervention)
  Change in cardiorespiratory fitness defined as the VO2peak obtained during a graded exercise test on a stationary bicycle.
Physical Function: Change in maximal knee extensor muscle power | 0 (pre-intervention) and 24 weeks (post-intervention)
  Change in maximal knee extensor muscle power obtained using dynamometry
Physical Function: Change in maximal knee extensor muscle strength | 0 (pre-intervention) and 24 weeks (post-intervention)
  Change in maximal knee extensor muscle strength assessed by one repetition maximum (1-RM)
Cognitive Function: Change in memory | 0 (pre-intervention) and 24 weeks (post-intervention)
  Change in memory will be measured using the Montreal Cognitive Assessment (MoCA Test). Max score of 30. Score of 26 and above is considered normal.
Cognitive Function: Change in learning | 0 (pre-intervention) and 24 weeks (post-intervention)
  Change in learning via the California Verbal Learning Test-III: learning slope for trials 1-5 and long delay retention (score range 0-16, where higher scores are better).
Cognitive Function: Change in executive function | 0 (pre-intervention) and 24 weeks (post-intervention)
  Change in executive function will be measured using the Executive function as indexed by: the Delis-Kaplan Executive Function System Trails Test, and Color-Word Interference Test (score range 0-19, where higher scores are better).
Metabolic Function: Change in hepatic insulin sensitivity | 0 (pre-intervention) and 24 weeks (post-intervention)
  Change in hepatic insulin sensitivity as assessed by suppression of endogenous glucose production during the dual tracer, 75g oral glucose tolerance test (OGTT)
Metabolic Function: Change in glucose variability | 0 (pre-intervention), 12, and 24 weeks (post-intervention)
  Glucose Variability will be assessed via continuous glucose monitoring during three occasions during weeks 0, 12, and 24 by measuring the change in range, total standard deviation, mean daily differences (MODD), and the overall net glycemic action over a 4-h and 8-h period (CONGA4; CONGA8).
Metabolic Function: Change in estimates of fasting insulin resistance | 0 (pre-intervention) and 24 weeks (post-intervention)
  Change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Metabolic Function: Change in whole body insulin sensitivity. | 0 (pre-intervention) and 24 weeks (post-intervention)
  Change in Matsuda Index where a higher value indicates greater insulin sensitivity
Metabolic Function: Change in insulin sensitivity and glucose clearance | 0 (pre-intervention) and 24 weeks (post-intervention)
  Change in oral glucose insulin sensitivity (OGIS) index where a higher value indicates greater insulin sensitivity
Change in whole blood DNA Methylated positions | 0 (pre-intervention) and 24 weeks (post-intervention)
  Change in differentially methylated positions in whole blood samples as assessed by whole-genome sequencing
Change in skeletal muscle transcriptome | 0 (pre-intervention) and 24 weeks (post-intervention)
  Transcriptomics: Change in skeletal muscle transcripts assessed via RNA sequencing
Change in concentration of lipid species | 0 (pre-intervention) and 24 weeks (post-intervention)
  Lipidomics: Change in the concentration of lipid species in blood and/or skeletal muscle as assessed by liquid chromatography mass spectrometry
Change in skeletal muscle protein abundance | 0 (pre-intervention) and 24 weeks (post-intervention)
  Proteomics: Change in abundance of skeletal muscle proteins as assessed by mass spectrometry.
Change in the concentration of metabolites | 0 (pre-intervention) and 24 weeks (post-intervention)
  Metabolomics: Change in concentration of blood and/or skeletal muscle metabolites as assessed by liquid chromatography mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Adam Konopka, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers years after the completion of the study endpoints by contacting Dr. Adam Konopka or the NIA BioBank Repository.